CLINICAL TRIAL: NCT01958528
Title: A Prospective Study Of Circulating Multiple Myeloma Cells As A Biomarker Of Progression In Myeloma Precursor States (MGUS And SMM)
Brief Title: Study Of Circulating Multiple Myeloma Cells As A Biomarker of MGUS And SMM
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 28412
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: a Diagnosis of MGUS or SMM by IMWG Criteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort 1 Progressors
- Cohort 2 - Non-Progressors

SUMMARY:
This is a prospective study to collect blood and bone marrow samples from patients with SM and MGUS. About 100 subjects will be enrolled at the University of Pennsylvania and followed for 2 years. The primary objective of this study is to evaluate CMMCs as a biomarker to detect patients at high risk of progression to multiple myeloma in patients with MGUS and SMM.

DETAILED DESCRIPTION:
The primary objective is to evaluate CMMCs as a biomarker to detect patients at high risk of progression to multiple myeloma in patients with MGUS and SMM. The secondary objective are to correlate CMMCs with the Mayo Clinic prognostic models in MGUS/SMM, to compare bone marrow genomic findings with genomic findings in CMMC (utilizing multiple myeloma FISH panel), to perform immunophenotyping of bone marrow plasma cells, to perform gene expression profiling on CD138+bone marrow plasma cells and correlate with progression, to perform serum microRNA profiling and correlate with progression, to correlate bone marrow immunohistochemical studies evaluating the microenvironment with CMMC, to perform proteomic profiling on peripheral blood to evaluate serum biomarkers of progression and to establish a biorepository of samples of peripheral blood for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Capable of informed consent
* A monoclonal gammopathy detected in the serum, including intact immunoglobulin (IgG and IgA) and light chain only gammopathies. Light chain only gammopathy is defined as an abnormal light chain ratio and increased involved light chain).44, 45
* Absence of myeloma related organ or tissue impairment ("CRAB") as defined by:

  * Hypercalcemia (calcium greater than or equal to 11)
  * Renal failure (creatinine >2.0)
  * Anemia hemoglobin <10 gm/dl)
  * Bone disease (Osteolytic lesions, fractures)

Exclusion Criteria:

* A secondary B-cell neoplasm or other active malignancy aside from non-melanoma skin cancer or localized prostate cancer. An active malignancy is any malignancy requiring therapy within the past 3 years. Patients with monoclonal B-cell lymphocytosis are not excluded.
* IgM monoclonal gammopathy
* Inability to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female subjects with diagnosis of MGUS or SMM by IMWG Criteria
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States